CLINICAL TRIAL: NCT05355376
Title: Colorectal Surgical Site Infection: a Cohort Study About How Can we Decrease it
Brief Title: Colorectal Surgical Site Infection
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar Universitário Lisboa Norte (Other)
Responsible Party: Principal Investigator, Aldara Filipa Peixoto Faria, Principal investigator, Centro Hospitalar Universitário Lisboa Norte
Other Study IDs: 0003
Record Dates: First submitted 2022-04-11; First posted 2022-05-02 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bundle of measures to decreased SSI

SUMMARY:
Surgical site infection (SSI) is one of the most common postoperative complications in surgery, with high morbidity. In the tertiary-center that the investigators evaluated they had a significant rate of surgical site infection. Because of that the investigators created a care bundle of measures in order to improve the outcomes.

DETAILED DESCRIPTION:
Prospectively the investigators implemented a care bundle of measures with retrospective analysis, to decrease SSI . The superficial, deep and organ/space infections were evaluated and compared before and after care bundle implementation.

Between january 1, 2016 and December 31, 2020, 1139 patient records relating to surgical incisions were submitted for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to elective colorectal surgery between 2016, january 1 and 2020, december 31
* Age > 18 years
* At least 30 days of follow-up

Exclusion Criteria:

* Patients submitted to urgent colorectal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to eletive colorectal surgery, by laparotomy, during a period of 5 years, in our colorectal department
Sampling Method: Non-Probability Sample
Enrollment: 1139 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
The rate of surgical site infections | 5 years
  Evaluate the variation of surgical site infections during a period of 5 years